CLINICAL TRIAL: NCT04707040
Title: Investigation of the Effects of Neurocognitive Exercise Program in Symptom Severity and Executive Functions in Children With Attention Deficit and Hyperactivity Disorder
Brief Title: Neurocognitive Exercise Program for Children With Attention Deficit and Hyperactivity Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dokuz Eylul University (Other)
Responsible Party: Principal Investigator, Ezgi Karagoz Tanigor M.D., Researcher, Dokuz Eylul University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ADHD-NEP
Record Dates: First submitted 2021-01-11; First posted 2021-01-13 (Actual); Last update posted 2021-01-20 (Actual); Status verified 2021-01

CONDITIONS: Attention Deficit Hyperactivity Disorder
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Masking Description: The investigator who performed the outcome measures were blind to the groups, and did not know if the participant was actually a healthy control, or a patient with ADHD.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Neurocognitive Exercise Program Group (Experimental): The group received NEP for 10 weeks, one hour per week conducted by the same physiotherapist with 6 years of experience in this field. Children with ADHD were given home exercises for the other six days of the week without a NEP session. Home exercises were followed with an exercise diary under the control of children's parents. The home exercise program consisted of visual-motor and auditory-motor coordination tasks (daily 15 min).
  Interventions: Other: Neurocognitive Exercise Program

INTERVENTIONS:
Other: Neurocognitive Exercise Program — Neurocognitive Exercise Program (NEP) is defined as a multimodal exercise program including different motor coordination exercises and cognitive tasks. Exercise progression is performed from easy to difficult, and consist of simple and complex tasks. Different sports equipment (such as different sizes of balls, racket, tulle, pilates ball, eye band, rope, etc.) is used in motor coordination exercises where multiple extremities can be used in NEP. These materials are used during different exercises including cross-limb movements, throwing, jumping, walking, involving different cognitive tasks. The cognitive task used and the degree of difficulty of the task are provided by different visual (colored cards, numbered cards, gestures, etc.) or auditory (keywords, ring signal, etc.) signs. For example, showing a red card might indicate throwing a ball with the left hand, while showing a blue card indicates throwing a ball with the right hand and walking forward

SUMMARY:
The effects of Neurocognitive Exercise Program (NEP) on ADHD symptoms and executive functions in children with Attention Deficit and Hyperactivity Disorder (ADHD) will be investigated using The Conners parent rating scale-revised short (CPRS-RS), Stroop Test, Wisconsin test and Y-Balance test.

DETAILED DESCRIPTION:
The effects of Neurocognitive Exercise Program (NEP) on ADHD symptoms and executive functions in children with Attention Deficit and Hyperactivity Disorder (ADHD) will be investigated.

Material and Methods: Twenty-nine boys (14 ADHD, 15 Healthy Controls) between 7 and 13 years of age will be recruited in the study and The Conners parent rating scale-revised short (CPRS-RS), Stroop Test, Wisconsin test and Y-Balance test will be performed . All tests and measurements will be performed for ADHD group before NEP, after NEP, 6 months and 12 months. The control group will be evaluated only once.

ELIGIBILITY:
Inclusion Criteria:

* Children between 7-13 years old
* Diagnosis of ADHD given by an experienced child psychiatrist based on the 5th edition of Diagnostic and Statistical Manual of Mental Disorders (American Psychiatric Association, 2013)

Exclusion Criteria:

* Presence of anxiety,
* Presence of depression,
* Presence of learning disability,
* Presence of intellectual disability,
* Presence of visual impairment,
* Presence of musculoskeletal or neurological disorders that may directly affect motor skill and cognition

Ages: 7 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 14 (Actual)
Dates: Start 2018-01-08 (Actual); Primary Completion 2020-01-08 (Actual); Study Completion 2020-01-08 (Actual)

PRIMARY OUTCOMES:
Stroop color-word test | 12 months
  The Stroop Color-Word Test is a color-word task assessing executive function involving processing speed, concentration, and attention (Stroop, 1935). Stroop Test was applied in five sections. These sections and related cards are as follows in their application order: (1) The card with the color names printed in black (1st card), (2) the card with the color names printed in different colors (2nd card), (3) the card with the colored printed circles (3rd card), (4) in the card with neutral words without the color name (4th Card), (5) The section where the colors of the words in the 2nd Card are spelled, with the names of colors printed in different colors. Stroop test gives information about many cognitive processes such as selective attention, focused attention, response inhibition, interference control, and information processing speed.
Conners parent rating scale-revised short (CPRS-RS) | 12 months
  CPRS-RS is a 27-item scale that determines the severity of ADHD. The items consist of three sub-scales (Disagree-QA, Cognitive Problems-Inattention CP-I, Hyperactivity-HI) and an auxiliary scale (ADHD Index). The questions are answered by the parents on a four-point Likert scale. "Never", "rarely", "often" and "always" options are scored as "0", "1", "2" and "3" respectively

SECONDARY OUTCOMES:
Wisconsin Card Sorting Test (WCST) | 12 months
  The WCST is a test used for executive function assessment, which includes measurements related to strategic planning, updating, shift cognitive set, modulating impulsive responding, and perseveration (Greve et al., 2005). The computer version of the test was used in this study (Heaton, 2008). The WCST included four stimulus cards and 128 response cards. Respondents were required to sort response cards based on one of three characteristics (i.e., color, form, and number) of the four stimulus cards. The computer gives 'correct' or 'wrong' feedback after each response. The ranking category changes when the participant selects the appropriate card for 10 cards. The test is completed after the participant has completed 6 categories or at the end of 128 response cards.
Y-Balance test | 12 months
  Y-Balance Test (YBT) was used to evaluate the dynamic balance of children. YBT was performed in three directions (anterior, posteromedial, and posterolateral). The test protocol was applied based on the learning effect (Hertel et al., 2000). After measuring the leg length (anterior superior iliac spine to the medial malleolus) of the children, the average of three measurements taken after 6 attempts in both directions with both feet was taken as the test score. [YBT normalized value: (Average of 3 reach distances) / limb length x 100; YBT composite score: (Anterior + Posteromedial + Posterolateral) / (3 x Limb Length) x100)].

CONTACTS AND LOCATIONS:
Overall Officials: Aylin Ozbek, MD, Principal Investigator — Dokuz Eylul University
Locations (1):
- Dokuz Eylul University, Izmir, Narlıdere, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chambers WJ, Puig-Antich J, Hirsch M, Paez P, Ambrosini PJ, Tabrizi MA, Davies M. The assessment of affective disorders in children and adolescents by semistructured interview. Test-retest reliability of the schedule for affective disorders and schizophrenia for school-age children, present episode version. Arch Gen Psychiatry. 1985 Jul;42(7):696-702. doi: 10.1001/archpsyc.1985.01790300064008. PMID 4015311
- [Background] Christiansen L, Beck MM, Bilenberg N, Wienecke J, Astrup A, Lundbye-Jensen J. Effects of Exercise on Cognitive Performance in Children and Adolescents with ADHD: Potential Mechanisms and Evidence-based Recommendations. J Clin Med. 2019 Jun 12;8(6):841. doi: 10.3390/jcm8060841. PMID 31212854
- [Background] Diedrichsen J, Criscimagna-Hemminger SE, Shadmehr R. Dissociating timing and coordination as functions of the cerebellum. J Neurosci. 2007 Jun 6;27(23):6291-301. doi: 10.1523/JNEUROSCI.0061-07.2007. PMID 17554003
- [Background] Goetz M, Schwabova JP, Hlavka Z, Ptacek R, Surman CB. Dynamic balance in children with attention-deficit hyperactivity disorder and its relationship with cognitive functions and cerebellum. Neuropsychiatr Dis Treat. 2017 Mar 21;13:873-880. doi: 10.2147/NDT.S125169. eCollection 2017. PMID 28356743
- [Background] Greve KW, Ingram F, Bianchini KJ. Latent structure of the Wisconsin Card Sorting Test in a clinical sample. Arch Clin Neuropsychol. 1998 Oct;13(7):597-609. PMID 14590620
- [Background] Kaufman J, Birmaher B, Brent D, Rao U, Flynn C, Moreci P, Williamson D, Ryan N. Schedule for Affective Disorders and Schizophrenia for School-Age Children-Present and Lifetime Version (K-SADS-PL): initial reliability and validity data. J Am Acad Child Adolesc Psychiatry. 1997 Jul;36(7):980-8. doi: 10.1097/00004583-199707000-00021. PMID 9204677
- [Background] Polanczyk G, de Lima MS, Horta BL, Biederman J, Rohde LA. The worldwide prevalence of ADHD: a systematic review and metaregression analysis. Am J Psychiatry. 2007 Jun;164(6):942-8. doi: 10.1176/ajp.2007.164.6.942. PMID 17541055
- [Background] Vysniauske R, Verburgh L, Oosterlaan J, Molendijk ML. The Effects of Physical Exercise on Functional Outcomes in the Treatment of ADHD: A Meta-Analysis. J Atten Disord. 2020 Mar;24(5):644-654. doi: 10.1177/1087054715627489. Epub 2016 Feb 9. PMID 26861158
- [Derived] Buker N, Karagoz E, Sengul YS, Guney SA, Ozbek A. Neurocognitive training enhances the outcomes of children with attention deficit hyperactivity disorder: A preliminary study. Child Care Health Dev. 2024 May;50(3):e13268. doi: 10.1111/cch.13268. PMID 38767513